CLINICAL TRIAL: NCT06195046
Title: Baroreflex Activation Therapy in Left Ventricular Assist Device Patients Study (BAT-VAD Study)
Brief Title: Baroreflex Activation Therapy in Left Ventricular Assist Device Patients Study
Acronym: BAT-VAD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not moving forward due to unable to identify patients who qualify.
Sponsor: Medical University of South Carolina (Other)
Collaborators: CVRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pro00115552
Record Dates: First submitted 2023-07-21; First posted 2024-01-08 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Congestive Heart Failure
Keywords: Ventricular Assist Device; Baroreflex activation therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: double-blind cross-over study design
Who Masked: Participant, Investigator
Masking Description: patient and Investigator will not know whether the subject has BAT turned on or off during each of the 3 month follow-up intervals
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- control (BAT off) (Sham Comparator): Baroreflex activation therapy turned off for three months
  Interventions: Device: Baroreflex Activation Therapy (BAT)
- treatment (BAT on) (Experimental): Baroreflex activation therapy turned on for three months
  Interventions: Device: Baroreflex Activation Therapy (BAT)

INTERVENTIONS:
Device: Baroreflex Activation Therapy (BAT) — activation of BAROSTIM NEO system that affects autonomic modulation with BAT therapy.

SUMMARY:
This study will involve LVAD patients who have already received a clinically-indicated BAT (BAROSTIM) device. After recovery from LVAD implant, we will investigate the effects of BAT in a double-blind cross-over study design.

DETAILED DESCRIPTION:
Left ventricular assist devices (LVADs) provide a meaningful therapeutic option for patients with end-stage systolic heart failure who cannot receive cardiac transplantation. For these patients, LVADs have been shown to improve mortality, functional capacity, and quality of life [1-3]. With ever-improving technological and procedural advances, the number of LVAD implantations for patients with end-stage cardiomyopathy as bridge to transplant, recovery, or even as destination therapy continues to rise [4]. Despite the short term clinical benefits of LVAD support, studies show that deleterious neurohormonal activation does not abate after LVAD implantation and that left ventricular scarring (or fibrosis) does not regress and may worsen. Similarly, the prevalence of myocardial recovery with LVAD support has been dismally low with <1% of patients recovering to the point where their LVAD can be safely explanted. Given that the majority of patients undergoing LVAD are now doing so with a destination therapy designation, and that the median estimated survival time on LVAD support ranges from 4-6 years, the importance of therapies to maximize chances for myocardial recovery while LVAD supported is evident.

The pathophysiologic reasons underlying the lack of abrogation of sympathetic and neurohormonal signaling with LVAD support, even in the face of adequate hemodynamic support, may center around the non-pulsatile nature of the device. Markham and Levine described sympathetic nerve activity in both pulsatile and nonpuslatile LVAD patients in 2013, demonstrating that patients with nonpulsatile devices had markedly elevated muscle sympathetic nerve activity, though pulsatile LVAD patients and normal controls had similar sympathetic activity. In a sequence of experiments, the authors demonstrated that this was at least partly due to baroreceptor unloading in the nonpulsatile patients. Further studies have demonstrated that plasma norepinephrine levels remain elevated after VAD implant, as do neurohormones in the renin-angiotensin-aldosterone axis. Sympathetic neurohormone levels have been shown to correlate with clinical response to LVAD therapy (defined by significant improvement in quality of life determined by the KCCQ), with reduced B-adrenergic receptor kinase-1 and DHPG levels differentiating those with better clinical response. Further, pathologic studies pre- and post-LVAD have demonstrated an acceleration of deleterious myocardial fibrosis during LVAD support, potentially driven by sympathetic and/or RAAS signaling pathways.

As demonstrated in preclinical studies and the clinical BeAT-HF trial, autonomic modulation with baroreflex activation therapy (BAT) with the BAROSTIM NEO system reduced sympathetic signaling, leading to increased NT-proBNP, 6-minute hall walk distance (6MHW), and improved quality of life in patients with chronic systolic heart failure.

However, the role of BAT in the unique physiologic LVAD-supported state has not be characterized. Given the concerns that LVAD support by augment sympathetic and thereby RAAS signaling, and that BAT may abrogate those deleterious pathways, we propose to study the clinical and neurohormonal effects of BAT in LVAD supported patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* LVAD patient > 3 months post implant
* Existing BAT device

Exclusion Criteria:

* Presence of cardiogenic shock, respiratory failure, hypotension or unstable heart failure
* Bradycardia (resting HR <60 beats/minute)
* Presence of suspected pump thrombosis at the time of enrollment
* Presence of any significant ventricular arrhythmias at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
6 Minute Hall Walk | 3 months
  change in distance walked during 6 Minute Hall Walk

SECONDARY OUTCOMES:
Minnesota Living with Heart Failure Questionnaire | 3 months, 6 months
  quality of life questionnaire
Change in LVAD system monitor reported flow | 3 months, 6 months
  Liters/minute
Cardiac 123-mIBG scan | 3 months, 6 months
  Heart to mediastinum uptake ratio; Rate of 123-mIBG washout
Change in left ventricular size on transthoracic echocardiogram | 3 months, 6 months
  Centimeters
Change in aortic valve opening frequency on transthoracic echocardiogram | 3 months, 6 months
  Valve opening per beat
Change in mitral valve regurgitation severity on transthoracic echocardiogram | 3 months, 6 months
  None, mild, moderate, severe
Change in right ventricular size on transthoracic echocardiogram | 3 months, 6 months
  Centimeters
Change in Serum catecholamines | 3 months, 6 months
  pg/mL
Change in Serum norepinephrine | 3 months, 6 months
  pg/mL
Change in serum renin | 3 months, 6 months
  ng/mL
Change in serum aldosterone | 3 months, 6 months
  ng/dL
Change in serum angiotensin | 3 months, 6 months
  U/L
Change in serum BNP | 3 months, 6 months
  pg/mL

IPD SHARING:
Plan to Share IPD: No